CLINICAL TRIAL: NCT03197675
Title: The Use of Acupuncture in Potentiating Functional Recovery in Spinal Cord Injury Subjects
Brief Title: Acupuncture in Spinal Cord Injury Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Deborah Stein, Chief of Trauma, Medical Director, Neurotrauma Critical Care, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00074616
Record Dates: First submitted 2017-06-19; First posted 2017-06-23 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Spinal Cord Injuries
Keywords: Chronic pain; Acupuncture
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Participants who are randomized to the control group will not receive any acupuncture. Participants will however be assessed weekly to obtain the same data on their pain scale and other outcome measures as the treatment group. Participants will be evaluated in person during their standard of care clinical follow up appointments at the three month and six month points for in person interviews and data collection .
  Interventions: Other: Acupuncture
- treatment group (Active Comparator): Participants within the acupuncture treatment group will receive traditional body acupuncture with electrical stimulation for 30 minutes three times a week, additionally participants will also receive auricular acupuncture once a week with the needles retained in both ears for seven days and replaced the following week, for a total of eight weeks (24 treatments of conventional acupuncture, 8 treatments of auricular acupuncture). Pain Numeric Rating Score (NRS) will be evaluated by the research staff before and after each treatment. All participants will then be reevaluated with the described assessment tools at three months and again at six months. Acupuncturists will not participate in the three and six month evaluations of subjects.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Participants within the acupuncture treatment group will receive traditional body acupuncture with electrical stimulation for 30 minutes three times a week, additionally participants will also receive auricular acupuncture once a week with the needles retained in both ears for seven days and replaced the following week, for a total of eight weeks (24 treatments of conventional acupuncture and 8 treatments of auricular acupuncture). Relative pain levels will be measured via the NRS by a member of the research staff before and after each treatment. All participants will then be reevaluated with the described assessment tools at three months and again at six months. Acupuncturists will not participate in the three and six month evaluations of subjects.

SUMMARY:
Of the more than 250,000 Americans with severe spinal cord injury (SCI), 42,000 are military veterans. The Department of Veterans Affairs is the largest single network of SCI care providers in the nation. Patients with SCI experience functional disabilities as well as chronic pain. Studies show that individuals with SCI report pain refractory to conventional treatments. Civilian and veteran patients with SCI have associated pain with impairments in physical and cognitive function, sleep, employment, social relationships, community re-integration and quality of life. In a survey of individuals with SCI, those who used acupuncture experienced a reduction of pain symptoms lasting hours after treatment, with 27.3% reporting pain relief for days. A pilot study on the use of auricular acupuncture for neuropathic pain associated with SCI showed a greater reduction of pain as measured by the Numerical Rating Scale (NRS). A recent review of randomized controlled trials regarding the use of acupuncture in SCI found that only two of sixteen included studies were of high quality. There was limited evidence for the use of acupuncture in motor functional recovery, bladder function recovery, and in pain control related to SCI. Further high quality studies are needed. This proposal is for a phase II randomized clinical trial.

DETAILED DESCRIPTION:
Objective/Hypothesis:

Our overarching hypothesis is that acupuncture is beneficial following acute traumatic SCI with respect to severity of neuropathic pain syndromes, patient-perceived quality of life measures, and functional outcomes. The current literature suggests that acupuncture may improve upon traditional pharmacological treatment results for SCI related pain, and that patients are seeking improved pain management in order to improve their quality of life. While data is limited, there may also be improvement in motor functional recovery with the use of acupuncture. We do know that SCI related pain limits patient participation in rehabilitation, thus advances in the management of SCI related pain is a priority in SCI research in order to improve outcomes after SCI.

Specific Aims:

Specific Aim 1: To determine whether patients treated with acupuncture started during acute care have better immediate and long-term pain scores and decreases in self-reported pain interference.

Specific Aim 2: To determine whether patients treated with acupuncture started during acute care will have better overall quality of life measurements and improvements in self-reported well-being and resilience.

Specific Aim 3: To determine whether patients treated with acupuncture started during acute care will have improvement in functional recovery in comparison to the control group.

Study Design:

This trial will compare pain scores and patient-perceived quality of life for individuals who receive early and regular acupuncture therapy to a control group. Patients with blunt or penetrating traumatic SCI will be included. The Investigators will enroll 100 subjects over a 36-month period from the R Adams Cowley Shock Trauma Center (STC). Once consent is obtained, enrolled patients will be evaluated using the ISNCSCI examination. Information about neuropathic pain and quality of life will be scored using NIH CDE recommended validated instruments within 72 hours of injury, during the 8-week treatment period, and at 3 and 6 months. The primary outcome is the improvement in NRS. The secondary outcomes are improvements in quality of life and functional recovery. Statistical analyses will involve constructive repeated measures mixed models to estimate the effect of treatment.

Clinical Impact:

The proposed trial will investigate the promising intervention of acupuncture for the management of neuropathic pain related to SCI. Improvement in neuropathic pain management is crucial in improving patients' rehabilitation, quality of life and ultimate outcome.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 75
2. complete (AIS A) or incomplete SCI (AIS B-D) of the cervical, thoracic or lumbar spine from blunt or penetrating trauma
3. ability to understand verbal and written English

Exclusion Criteria:

1. a history of peripheral neuropathy
2. medical diagnoses or conditions that preclude them from active participation (for example, moderate or severe traumatic brain injury)
3. receipt of acupuncture in the last three months prior to enrollment
4. presence of skin breakdown or infection over the extremities or external ears
5. active participation in other research studies
6. cognitive impairment that prevents understanding the test instructions
7. prisoner
8. pregnancy
9. active duty military personnel
10. individuals who do not speak or understand the English language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Compare pain assessments in patients with SCI treated with acupuncture to patients treated per standard of care alone to assess for efficacy and durability of the effect on pain following SCI. | within 3 months following hospital discharge
  All enrolled patients will be evaluated using the complete ISNCSCI examination. Information about neuropathic pain will be scored using the ISCIPBDS (version 2.0) and ISCIPEDS. A SCI-QOL will be administered during the three month reevaluations to assess the patient's perceived quality of life. In the intervening weeks a select few ISCIPBDS items will be administered on a weekly basis until study completion.

SECONDARY OUTCOMES:
Compare pain assessments in patients with SCI treated with acupuncture to patients treated per standard of care alone to assess for efficacy and durability of the effect on pain following SCI. | within 6 months following hospital discharge
  All enrolled patients will be evaluated using the complete ISNCSCI examination. Information about neuropathic pain will be scored using the ISCIPBDS (version 2.0) and ISCIPEDS. A SCI-QOL will be administered during the six month reevaluations to assess the patient's perceived quality of life. In the intervening weeks a select few ISCIPBDS items will be administered on a weekly basis until study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Stein, MD, MPH, Principal Investigator — Professor of Surgery, Department of Surgery, Chief of Trauma R Adams Cowley Shock Trauma Center
Locations (1):
- R Adams Cowley Shock Trauma Center, University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No